CLINICAL TRIAL: NCT06630897
Title: Art and Science of Human Flourishing Microsupport Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-0929; A171600 (Other: UW Madison); Protocol Version 10/21/24 (Other: UW Madison)
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Mental Stress
Keywords: Wellbeing; Digital Support; Microsupport; text messages
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Microsupport (Experimental)
  Interventions: Other: Text Messages
- No Microsupport (No Intervention)

INTERVENTIONS:
Other: Text Messages — small amounts of digital support will be in the form of text messages
  Arms: Microsupport

SUMMARY:
The purpose of this study is to determine whether providing small amounts of digital support impacts students in the Art and Science of Human Flourishing (ASHF) course. Approximately 300 participants will be enrolled and can expect to be on study for up to 4 months.

DETAILED DESCRIPTION:
Participants will be currently enrolled students in the ASHF course. Students will complete measures at baseline, daily during the 1-month intervention period, at post-treatment, and 3 months later. During the 1-month intervention period, half of the participants will be randomized to receive small amounts of digital support in the form of text messages.

Context (from the course website): The Art and Science of Human Flourishing course is taught in tandem with the Healthy Minds Program (HMP) app. The overall framework of the ASHF course largely aligns with the HMP app and is composed of the following modules and sub-themes which are covered throughout the course of a 15-week semester:

Foundations: Flourishing, Transformation, Resilience

* Awareness: Focus, Emotions, Mindfulness
* Connection: Interdependence, Compassion, Diversity
* Wisdom: Identity, Values, Gratitude
* Integration: Courage, Community

Small amounts of digital support will be tested on half the participants. Primary Outcomes for measuring the effect of this support will be the PROMIS Depression and Anxiety Measures.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in ASHF course

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Daily Informal Practice | Data collected each evening throughout the intervention (up to 1 month)
  Daily informal practice will be measured by a single item: "Today, I have tried to apply the practices I have been learning in the HMP app to my day-to-day activities." Participants will respond on a Likert scale (1 = not at all, 5 = all day long). A higher score on this item indicates more informal practice on that day.
Daily psychological distress | Data collected each evening throughout the intervention (up to 1 month)
  Daily psychological distress will be measured by two items on anxiety ("Today, I felt anxious") and depression ("Today, I felt depressed"). Participants will rate these items on a 5-point Likert scale (1 = not at all, 5 = very much). Responses to each item will be z-scored and then averaged to create a distress composite.

SECONDARY OUTCOMES:
Composite Psychological Distress Score | baseline, 1 month (immediately post-intervention), 4 months (3 month post-intervention follow up)
  A composite psychological distress score will be obtained by computing a mean across scaled (z-transformed) scores on the computer-adaptive versions of PROMIS Depression and PROMIS Anxiety Scales and NIH Toolbox 10-item Perceived Stress. For PROMIS Depression Scale, participants score 4 to 8 items on a 5 point Likert scale from 1 (never) to 5 (always) to measure how they felt in the past 7 days. For PROMIS Anxiety Scale, participants score 4 to 8 items on a 5 point Likert scale from 1 (never) to 5 (always) to measure how they felt in the past 7 days. For NIH Toolbox 10-item Perceived Stress, participants score on a 5 point Likert scale from 1 (never) to 5 (very often) to measure how they felt in the past 7 days.
NIH Toolbox Loneliness Score | baseline, 1 month (immediately post-intervention), 4 months (3 month post-intervention follow up)
  5-item survey scored from 1 (never) to 5 (always), where higher overall scores indicate higher loneliness.
PROMIS Sleep Disturbance Score | baseline, 1 month (immediately post-intervention), 4 months (3 month post-intervention follow up)
  The computer adaptive version will draw from a bank of 27-items scored from 1 (never / very poor) to 5 (always / very good), where higher overall scores indicate greater sleep disturbance in the past 7 days.
Drexel Defusion Scale score | baseline, 1 month (immediately post-intervention), 4 months (3 month post-intervention follow up)
  10-item survey scored from 0 (not at all) to 5 (very much), where higher overall scores indicate higher defusion.
Experiences Questionnaire Decentering Score | baseline, 1 month (immediately post-intervention), 4 months (3 month post-intervention follow up)
  11-item survey scored from 1 (never) to 5 (all the time), where higher overall scores indicate higher levels of decentering.
Sense of Belonging Score | baseline, 1 month (immediately post-intervention), 4 months (3 month post-intervention follow up)
  8-item survey scored from 1 (not at all true for me) to 5 (very true for me), where higher overall scores indicate higher sense of belonging.
Five Facet Mindfulness Questionnaire Awareness Subscale Score | baseline, 1 month (immediately post-intervention), 4 months (3 month post-intervention follow up)
  8-item survey scored from 1 (never or very rarely true) to 5 (very often or always true) where higher overall scores indicate higher awareness.
Healthy Minds Index Scores | baseline, 1 month (immediately post-intervention), 4 months (3 month post-intervention follow up)
  17-item survey scored from 0 (not at all / never / none of the time) to 4 (to the highest degree / always / all of the time) on each of 4 domains: Awareness, Connection, Insight, Purpose. Higher overall scores indicate higher sense of awareness, connection, insight, and purpose.
Digital Working Alliance Inventory (D-WAI) Score | 1 month (immediately post-intervention), 4 months (3 month post-intervention follow up)
  6-item survey scored from 1 (strongly disagree) to 7 (strongly agree), where higher overall scores indicate higher digital working alliance.
Mindfulness Adherence Questionnaire Score | 1 month (immediately post-intervention), 4 months (3 month post-intervention follow up)
  10-item survey scored from 0 (never) to 6 (always), where higher overall scores indicate higher quality of mindfulness practice. A four-item subscale can be computed for formal practice and a six-item subscale can be computed for informal practice.
Alcohol Use Disorders Identification Test Score | baseline, 1 month (immediately post-intervention), 4 months (3 month post-intervention follow up)
  10-item survey scored from 0 (never / no / 1 or 2) to 4 (4 or more times a week / 10 or more / daily or almost daily / yes, during the past year). Higher overall scores indicate higher alcohol use concerns.
Morning mindfulness, decentering, connection, purpose, depression, anxiety, stress, rumination, and motivation to practice scores | Each morning throughout the intervention (up to 1 month)
  Morning mindfulness, decentering, connection, purpose, depression, anxiety, stress, rumination, and motivation to practice meditation will be measured by a single item, respectively. Participants will respond on a Likert scale (1 = not at all, 5 = very much). A higher score on these items indicates higher mindfulness, decentering, loneliness, purpose, depression, anxiety, stress, rumination, sleep quality, and motivation to practice meditation that morning.
Sleep quality scores | Each morning throughout the intervention (up to 1 month)
  For sleep quality, participants will respond on a Likert scale (1 = very bad, 4 = very good). A higher score indicates better sleep quality.
Evening mindfulness, decentering, connection, purpose, happy event, stressor exposure, rumination scoring | Each evening throughout the intervention (up to 1 month)
  Evening mindfulness, decentering, connection, purpose, happy event, stressor exposure, rumination, and formal practice will be measured by a single item, respectively. Participants will respond on a Likert scale (1 = not at all, 5 = very much). A higher score on the items indicates higher mindfulness, decentering, loneliness, purpose, happiness, stress, and rumination that day.
Percentage of Participants with a formal practice | Each evening throughout the intervention (up to 1 month)
  Participants will respond yes or no to whether they have a mindfulness, decentering, connection, purpose, happy event, stressor exposure, rumination formal practice. A response of "Yes" to the formal practice item indicates that the participant used the HMP app on that day, while a response of "No" indicates non-use.
Acceptability of Intervention Measure Score | 1 month (immediately post-intervention)
  The Acceptability of Intervention Measure is a 4-item self-report measure scored on a 5-point likert scale from 1 (completely disagree) to 5 (completely agree), where higher scores indicate greater acceptability of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Goldberg, PhD, Principal Investigator — Center for Healthy Minds
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Art and Science of Human Flourishing Course — https://centerhealthyminds.org/the-art-and-science-of-human-flourishing-course

DOCUMENTS (1):
  • Informed Consent Form (2024-09-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT06630897/ICF_000.pdf